CLINICAL TRIAL: NCT04748666
Title: Problem Solving Training (PST) for English- and Spanish-speaking Care Partners of Adults With Alzheimer's and Alzheimer'S-related Dementia
Brief Title: PST for Care Partners of Adults With Alzheimer's and Alzheimer'S-related Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: University of Texas Rio Grande Valley (Other); Texas A&M University (Other)
Responsible Party: Principal Investigator, Shannon Juengst, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: STU-2020-1276
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Alzheimer Disease; Frontotemporal Degeneration (FTD); Lewy Body Dementia (LBD); Vascular Contributions to Cognitive Impairment and Dementia (VCID); Mixed Etiology Dementias (MED); Mild Cognitive Impairment (MCI)
Keywords: Alzheimer Disease; Frontotemporal Degeneration; Lewy Body Dementia; Vascular contributions to cognitive impairment and dementia; Mixed etiology dementias; Mild Cognitive Impairment; Care partner; Caregiver; Alzheimer's-related Dementia
MeSH Terms: conditions — Alzheimer Disease; Lewy Body Disease; Dementia; Mixed Dementias; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: The investigators will compare a) care partner emotional symptom (depression) change and b) caregiver burden change from baseline to 6-months post-baseline, to assessed long-term effects of PST and booster sessions several months beyond completion of the training. The investigators will also measure secondary care partner outcomes, including caregiver self-efficacy, positive aspects of caregiving, and alcohol use. Finally, the investigators will assess care partners' satisfaction, confidence using the PST strategy, and engagement across all conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 3 PST sessions and no boosters (Experimental)
  Interventions: Behavioral: Problem Solving Training
- 3 PST sessions with monthly boosters for 6 months (Experimental)
  Interventions: Behavioral: Problem Solving Training
- 6 PST sessions, no boosters (Experimental)
  Interventions: Behavioral: Problem Solving Training
- 6 PST sessions with monthly boosters for 6 months (Experimental)
  Interventions: Behavioral: Problem Solving Training

INTERVENTIONS:
Behavioral: Problem Solving Training — Problem Solving Training (PST) is a metacognitive strategy training approach, grounded in self-management theory, that teaches a simple, systematic method for evaluating problems, generating and selecting solutions, developing specific goals and action plans, and evaluating and revising plans as needed.

SUMMARY:
Caregivers of individuals with Alzheimer's disease and related dementia rarely get the preparation or training they need to manage their caregiving responsibilities and to successfully balance their own self-care and their caregiving roles. As a result, caregivers often experience caregiver burden, emotional distress, and substance abuse. Therefore, there is a critical need to support the emotional and social functioning of caregivers to improve their health and well-being and to prevent caregiver burden and poor coping.

Problem solving training (PST) is an evidence-based approach that teaches and empowers individuals to solve emergent problems contributing to their depressive symptoms, helps improve coping skills and increases self-efficacy. However, critical gaps in knowledge and care remain regarding the necessary components of training (eg. How many sessions? What is the influence of personal factors?) that affect how effective PST is for individual caregivers. Finally, caregiver interventions have almost exclusively been tested in English-speaking caregivers, further contributing to existing health disparities among minority groups.

To address this critical need, Dr. Shannon Juengst, Assistant Professor of Physical Medicine and Rehabilitation was awarded a new Texas Alzheimer's Research and Care Consortium Collaborative Research Grant entitled, "Problem Solving Training (PST) for English- and Spanish-speaking Care Partners of Adults with Alzheimer's and Alzheimer's Related Dementia." For this project, Dr. Juengst has assembled a strong, multidisciplinary team with Dr. Gladys Maestre, Professor of Biomedical Sciences and Director of the NIA funded-Alzheimer's Disease Resource Center for Minority and Aging Research and Memory Disorders Center at UT Rio Grande Valley and Dr. Matthew Smith, Associate Professor of Environmental and Occupational Health and Co-Director of the Center for Population Health and Aging at Texas A&M University.

This project will establish the necessary guidelines for an evidence-based, implementable problem-solving intervention for both English- and Spanish-speaking caregivers to improve their health and well-being and identify potential mechanisms of action for such training.

DETAILED DESCRIPTION:
Over 65 million people in the United States currently provide informal (i.e. unpaid) care to an individual with a chronic illness or disability,1 including the nearly 6 million adults currently living with Alzheimer's disease (AD).2 Care partners of adults with AD and related dementias (AD/ADRD) often experience high caregiver burden, leading to emotional distress, depression, problematic alcohol use, health problems, isolation, and poor quality of life.3,4 Interventions to reduce care partner stress may reverse the negative impact of caregiver burden.5 The Global Impact of Dementia 2013-2050 policy brief specifically called for better education and skills training for care partners. Therefore, there is a critical need to provide evidence-based support to care partners so they can best manage their own lives and their care recipients' chronic health conditions.6

Problem-Solving Training (PST) is an evidence-based metacognitive strategy training approach that teaches a simple, systematic method for evaluating problems, generating and selecting solutions, developing specific goals and action plans, and evaluating and revising plans as needed.7-18 Individuals learn to set achievable goals under the coaching of a therapist and gain self-efficacy as they begin to see that the seemingly overwhelming problems are indeed solvable when approached in a stepwise, rational fashion. Few care partner interventions include problem-solving skills training to translate knowledge into meaningful action, leaving care partners struggling to effectively manage their own lives and their caregiving responsibilities. Additionally, as of 2018 Hispanic individuals make up roughly 39.6% of the population of Texas,19 but most care partner intervention studies exclude Spanish-speaking participants. Our team has translated and culturally adapted PST specifically for Spanish-speaking care partners,20 presenting the opportunity to close a critical health disparity among care partners in Texas. PST, in both English and Spanish, could be incorporated across clinical settings into existing education-based care partner interventions to fill the current gaps in clinical practice. PST for fcare partners may also improve care recipient outcomes as well.

Our long-term goal is to improve the health, well-being, and participation of care partners and individuals with AD/ADRD. Our multidisciplinary team has expertise in AD/ADRD and in delivering and evaluating PST. The investigators represent a multi-site collaborative leveraging the broader TARCC network. Our expertise and strong clinical and research environments ensure the rigor, clinical relevance, and feasibility of our proposed research. The investigators will conduct a multi-site randomized controlled trial with a factorial design of PST for care partners of adults with AD/ADRD to address the following specific aims:

Aim 1: Determine the optimal number of Problem Solving Training (PST) sessions and boosters to improve emotional symptoms and burden in English and Spanish speaking care partners of adults with AD/ADRD.

Hypothesis: Six PST sessions vs three sessions will be optimal for improving emotional symptoms and burden of both English and Spanish speaking care partners 6 months after baseline.

Hypothesis: Monthly brief booster sessions vs no boosters will be optimal for improving emotional symptoms and burden of both English and Spanish speaking care partners 6 months after baseline.

The investigators will compare a) care partner emotional symptom (depression) change and b) caregiver burden change from baseline to 6-months post-baseline, to assessed long-term effects of PST and booster sessions several months beyond completion of the training. The investigators will also measure secondary care partner outcomes, including caregiver self-efficacy, positive aspects of caregiving, and alcohol use. Finally, the investigators will assess care partners' satisfaction, confidence using the PST strategy, and engagement across all conditions.

Aim 2: Identify factors associated with response to treatment.

Hypothesis: Response to treatment will be associated with age, gender, engagement in and uptake of PST, working alliance, and goal attainment. To test this hypothesis, the investigators will assess the extent to which each of these factors predicts response to PST (change in outcome) using multiple linear regression.

Establishing specific guidelines for an evidence-based, implementable problem-solving intervention for both English and Spanish speaking care partners will result in direct clinical application to improve care partner health and well-being and to improve care recipient health and quality of life. The investigators will explore potential mechanisms of change for future prospective study. This proposal directly aligns with the mission of TARCC to take novel and innovative approaches to increase participation of diverse and underserved populations, promote collaboration across TARCC institutions, and contribute to advancement in therapeutic interventions to improve the lives of individuals with AD and related dementias.

Design. The investigators will conduct a randomized control trial of PST for care partners of adults with AD/ADRD to assess the effects of number of sessions (3 vs 6) and brief telephone booster sessions (boosters vs no boosters) on depressive symptoms (Patient Health Questionnaire-9) and caregiver burden (Zarit Burden Interview). The investigators will recruit n=180 participants (n=45 per arm) across our two enrollment sites and conduct assessments at baseline, end of intervention, and 6-months post-baseline. Booster sessions will begin 1 month after completion of PST and will occur monthly thereafter up to 6-months post-baseline conditions.

Randomization and Allocation. Randomization will be stratified by language and gender, then will occur in blocks of 16 (i.e. 4 participants allocated to each of the 4 conditions within each block). The investigators will uniformly sample (i.e. equal probability) random numbers from a set containing four 1's, four 2's, four 3's, and four 4's to generate the randomization table within each block.

Data Analysis & Sample Size Determination: The investigators will conduct Bayesian mixed-effect ordered logistic regression models with subject-specific random effects to identify the optimal intervention group for our two primary outcomes at 6-months post-baseline (Aim 1). The investigators will apply the same statistical analysis approach to secondary outcome measures. The posterior probability that receiving 6-sessions decreases the odds ratio of higher PHQ-9 and ZBI scores and that receiving a booster decreases the odds ratio of higher PHQ-9 and ZBI scores will be reported in lieu of a p-value, which is inexistent in the Bayesian paradigm. In accordance with the approach used to power the current study, a significant result for any of the three treatments will be defined as a posterior probability greater than 98.33% in order to achieve an overall experiment-wise significance level of 5%. The investigators will apply the same statistical analysis approach to secondary care partner outcomes (caregiver self-efficacy, positive aspects of caregiving, coping, and alcohol use). To identify factors associated with PST response to intervention (Aim 2), the investigators will conduct the following exploratory analyses. Based on the PHQ-9 minimal clinically important difference (MCID) for individual change of 5 points,32 The investigators will categorize participants into one of three response to intervention groups: Response group (PHQ-9 score decrease by >5 points from baseline to 6-months), No Change group (PHQ-9 scores are within +5 points of baseline at 6-months), and Decliner group (PHQ-9 scores increase by >5 points at 6-months). The investigators will examine predictors of response to intervention group using multinomial logistic regression. The investigators will further explore predictors of change in primary and secondary outcomes from baseline to 6-months post-intervention using multiple linear regression.

Based on 1,000 iterations of a simulation of our pilot data (PST to improve PHQ-9 in care partners in a different clinical population14), the sample size necessary to detect a 30% decrease in the odds ratio for those who received six sessions or a 30% decrease in the odds ratio for those who received booster sessions with at most 5% significance level and at least 80% power was found to be 23 per arm (4 arms) per center (2) for a total of n=184 total (n=203 accounting for 10% attrition).

ELIGIBILITY:
Inclusion Criteria:

* PHQ2 Score of 2 or higher and/or ZBI4 Score of 2 or higher
* 18 years or older
* Able to speak fluently in English or Spanish
* Cognitively able to make decisions, as determined by ability to provide informed consent
* Care partner/caregiver to individual with AD/ADRD
* Individual must have at least one year or more of a relationship with patient with AD/ADRD

Exclusion Criteria:

* Dispute over care partner's role in the care of patient
* Has previously participated in other PST study at UTSW within the past year
* Does not meet all the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female, Male, Transgender/other
Enrollment: 94 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
The Mean Change in Patient Health Questionnaire (PHQ-8) Score | Baseline, 6 months
  Patient Health Questionnaire (PHQ-9) assesses DSIM-IV-TR symptoms that define major depressive episode. Scores range from 0-27 for severity. The PHQ8 omits the final question about suicidality, resulting in a validated scale with scores ranging from 0-24.: 0-4 (none), 5-9 (mild), 10-14 (moderate), 15-19 (moderately severe), and >20 (severe).
The Mean Change in Zarit Burden Interview Score | Baseline, 6 months
  Zarit Burden Interview (ZBI) is a 22-item self-reported measure of perceived caregiver burden, including items related to psychological and emotional health, well-being, social and family life, finances, and perceive control. Cutoff scores are mild: 2-20; mild to moderate: 21-40; moderate to severe:41-60; severe: 61-88 burden

SECONDARY OUTCOMES:
The Mean Change in Family Caregivers Scale/Caregiver experience Score | Baseline, 6 months
  The Family Caregiving Scale (also referred to as the Caregiving Experience Scale) measures multiple dimensions mentioned below in detail. Higher scores indicate more of that particular scale.
  * Emotional well-being and physical health
  * Scales: Life Satisfaction, Social Support, and Carer Overload (scores from 6- 20, 7-35, and 3-15, respectively).
  * Caring Role
  * Scales: Satisfaction, Resentment, and Anger (scores from 6-30, 5-25, and 4-20, respectively).
  * Behavioral Problems Scales: Aggressive, Depressive, and Forgetfulness/confusion (scores from 9-36, 4-16, and 5-20, respectively).
  * Help provided by recipient Scales: Personal ADL/Instrumental ADL (scores from 0-7 and 0-4, respectively).
  * Help provided by carer Scales: Personal ADL/Instrumental ADL (scores from 0-7 and 0-4, respectively).
  * Family environment Scales: Closeness/Conflict (scores from 3-9 and 3-9, respectively).
The Mean Change in Client Satisfaction Questionnaire (CSQ-8) Score | 6 months
  Client Satisfaction Questionnaire (CSQ-8) is an 8-item measure of an individual's satisfaction with health-related services they have received, yielding a single summed score (ranging from 8 to 32) measuring overall satisfaction . Higher scores indicating high satisfaction.
Upstream Social Isolation Risk Screener (U-SIRS13) | Baseline, 6 months
  The Upstream Social Isolation Risk Screener (U-SIRS) is a 13-item scale that measures an individuals' feelings of disconnectedness, which encompasses aspects of social isolation and loneliness. The U-SIRS-13 yields a single summed score (ranging from 0 to 13) measuring overall risk of being disconnected. Higher scores indicate higher risk.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Juengst, Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (3):
- United States (3):
  - Texas A&M University, College Station, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Rio Grande Valley, Edinburg, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brookmeyer R, Abdalla N, Kawas CH, Corrada MM. Forecasting the prevalence of preclinical and clinical Alzheimer's disease in the United States. Alzheimers Dement. 2018 Feb;14(2):121-129. doi: 10.1016/j.jalz.2017.10.009. Epub 2017 Dec 7. PMID 29233480
- [Background] Wolff JL, Spillman BC, Freedman VA, Kasper JD. A National Profile of Family and Unpaid Caregivers Who Assist Older Adults With Health Care Activities. JAMA Intern Med. 2016 Mar;176(3):372-9. doi: 10.1001/jamainternmed.2015.7664. PMID 26882031
- [Background] Rospenda KM, Minich LM, Milner LA, Richman JA. Caregiver burden and alcohol use in a community sample. J Addict Dis. 2010 Jul;29(3):314-24. doi: 10.1080/10550887.2010.489450. PMID 20635281
- [Background] Allen AP, Curran EA, Duggan A, Cryan JF, Chorcorain AN, Dinan TG, Molloy DW, Kearney PM, Clarke G. A systematic review of the psychobiological burden of informal caregiving for patients with dementia: Focus on cognitive and biological markers of chronic stress. Neurosci Biobehav Rev. 2017 Feb;73:123-164. doi: 10.1016/j.neubiorev.2016.12.006. Epub 2016 Dec 13. PMID 27986469
- [Background] Prince M, Guerchet M, Prina M. The Global Impact of Dementia 2013-2050. Alzheimer's Disease International; 2013.
- [Background] Rivera PA, Elliott TR, Berry JW, Grant JS. Problem-solving training for family caregivers of persons with traumatic brain injuries: a randomized controlled trial. Arch Phys Med Rehabil. 2008 May;89(5):931-41. doi: 10.1016/j.apmr.2007.12.032. PMID 18452743
- [Background] Powell JM, Fraser R, Brockway JA, Temkin N, Bell KR. A Telehealth Approach to Caregiver Self-Management Following Traumatic Brain Injury: A Randomized Controlled Trial. J Head Trauma Rehabil. 2016 May-Jun;31(3):180-90. doi: 10.1097/HTR.0000000000000167. PMID 26394294
- [Background] Pfeiffer K, Beische D, Hautzinger M, Berry JW, Wengert J, Hoffrichter R, Becker C, van Schayck R, Elliott TR. Telephone-based problem-solving intervention for family caregivers of stroke survivors: a randomized controlled trial. J Consult Clin Psychol. 2014 Aug;82(4):628-43. doi: 10.1037/a0036987. Epub 2014 Jun 9. PMID 24911421
- [Background] Elliott TR, Berry JW, Grant JS. Problem-solving training for family caregivers of women with disabilities: a randomized clinical trial. Behav Res Ther. 2009 Jul;47(7):548-58. doi: 10.1016/j.brat.2009.03.006. Epub 2009 Mar 24. PMID 19361781
- [Background] Elliott TR, Berry JW. Brief problem-solving training for family caregivers of persons with recent-onset spinal cord injuries: a randomized controlled trial. J Clin Psychol. 2009 Apr;65(4):406-22. doi: 10.1002/jclp.20527. PMID 19229946
- [Background] Elliott TR, Shewchuk RM, Scott J. Family caregiver social problem-solving abilities and adjustment during the inital year of the caregiving role. J Couns Psychol. 2001;48(2):223-232. doi:10.1037/0022-0167.48.2.223
- [Background] Juengst SB, Silva V, Goldin Y, Cicerone K, Lengenfelder J, Chiaravalloti N, Driver S, Mellick D, Dart G, Kew CL, Nabasny A, Bell KR. Care partner problem solving training (CP-PST) for care partners of adults with traumatic brain injury during inpatient rehabilitation: Study protocol for a multisite, randomized, single-blind clinical feasibility trial. Contemp Clin Trials. 2019 May;80:9-15. doi: 10.1016/j.cct.2019.03.004. Epub 2019 Mar 16. PMID 30885800
- [Background] Juengst SB, Osborne CL, Holavanahalli R, Silva V, Kew CL, Nabasny A, Bell KR. Feasibility Study of Problem-Solving Training for Care Partners of Adults With Traumatic Brain Injury, Spinal Cord Injury, Burn Injury, or Stroke During the Inpatient Hospital Stay. Arch Rehabil Res Clin Transl. 2019 Jun 27;1(3-4):100009. doi: 10.1016/j.arrct.2019.100009. eCollection 2019 Dec. PMID 33543049
- [Background] Garand L, Morse JQ, ChiaRebecca L, Barnes J, Dadebo V, Lopez OL, Dew MA. Problem-solving therapy reduces subjective burden levels in caregivers of family members with mild cognitive impairment or early-stage dementia: Secondary analysis of a randomized clinical trial. Int J Geriatr Psychiatry. 2019 Jul;34(7):957-965. doi: 10.1002/gps.5095. Epub 2019 Apr 17. PMID 30868641
- [Background] Chiu M, Pauley T, Wesson V, Pushpakumar D, Sadavoy J. Evaluation of a problem-solving (PS) techniques-based intervention for informal carers of patients with dementia receiving in-home care. Int Psychogeriatr. 2015 Jun;27(6):937-48. doi: 10.1017/S1041610214002798. Epub 2015 Jan 23. PMID 25615434
- [Background] Domingues NS, Verreault P, Hudon C. Reducing Burden for Caregivers of Older Adults With Mild Cognitive Impairment: A Systematic Review. Am J Alzheimers Dis Other Demen. 2018 Nov;33(7):401-414. doi: 10.1177/1533317518788151. Epub 2018 Jul 24. PMID 30041535
- [Background] Beinart N, Weinman J, Wade D, Brady R. Caregiver burden and psychoeducational interventions in Alzheimer's disease: a review. Dement Geriatr Cogn Dis Extra. 2012 Jan;2(1):638-48. doi: 10.1159/000345777. Epub 2012 Dec 15. PMID 23341829
- [Background] Vega M, Nabasny A, Juengst SB. "Descubriendo Soluciones Juntos"-An argument for adapting problem-solving training for Latinx care partners after traumatic brain injury (TBI). Rehabil Psychol. 2020 Nov;65(4):337-346. doi: 10.1037/rep0000310. Epub 2020 Jan 23. PMID 31971433
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Hébert R, Bravo G, Préville M. Reliability, Validity and Reference Values of the Zarit Burden Interview for Assessing Informal Caregivers of Community-Dwelling Older Persons with Dementia<a href=
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Gitlin LN, Roth DL, Burgio LD, Loewenstein DA, Winter L, Nichols L, Arguelles S, Corcoran M, Burns R, Martindale J. Caregiver appraisals of functional dependence in individuals with dementia and associated caregiver upset: psychometric properties of a new scale and response patterns by caregiver and care recipient characteristics. J Aging Health. 2005 Apr;17(2):148-71. doi: 10.1177/0898264304274184. PMID 15750049
- [Background] Clifford C, Greenfield TK. The UCSF Client Satisfaction Scales: I. The Client Satisfaction Questionnaire-8. In: The Use of Psychological Testing for Treatment Planning and Outcomes Assessment, 2nd Ed. Lawrence Erlbaum Associates Publishers; 1999:1333-1346.
- [Background] Tarlow BJ, Wisniewski SR, Belle SH, Rubert M, Ory MG, Gallagher-Thompson D. Positive Aspects of Caregiving: Contributions of the REACH Project to the Development of New Measures for Alzheimer's Caregiving. Res Aging. 2004;26(4):429-453. doi:10.1177/0164027504264493
- [Background] Steffen AM, McKibbin C, Zeiss AM, Gallagher-Thompson D, Bandura A. The revised scale for caregiving self-efficacy: reliability and validity studies. J Gerontol B Psychol Sci Soc Sci. 2002 Jan;57(1):P74-86. doi: 10.1093/geronb/57.1.p74. PMID 11773226
- [Background] Hatcher RL, Gillaspy JA. Development and validation of a revised short version of the Working Alliance Inventory. Psychother Res. 2006;16(1):12-25.
- [Background] Nezu AM, Nezu CM, D'Zurilla TJ. Solving Life's Problems. New York: Springer; 2007.
- [Background] Malouff JM, Thorsteinsson EB, Schutte NS. The efficacy of problem solving therapy in reducing mental and physical health problems: a meta-analysis. Clin Psychol Rev. 2007 Jan;27(1):46-57. doi: 10.1016/j.cpr.2005.12.005. Epub 2006 Feb 9. PMID 16480801
- [Background] Malec JF. Goal Attainment Scaling in Rehabilitation. Neuropsychol Rehabil. 1999;9(3-4):253-275. doi:10.1080/096020199389365
- [Background] Lowe B, Kroenke K, Grafe K. Detecting and monitoring depression with a two-item questionnaire (PHQ-2). J Psychosom Res. 2005 Feb;58(2):163-71. doi: 10.1016/j.jpsychores.2004.09.006. PMID 15820844
- [Derived] Juengst SB, Smith ML, Wilmoth K, Wright B, Han G, Supnet C, Maestre G. Problem-solving training to improve caregiver burden and depressive symptoms among dementia caregivers: personal and clinical factors of responders vs. non-responders. Front Public Health. 2025 Oct 10;13:1682373. doi: 10.3389/fpubh.2025.1682373. eCollection 2025. PMID 41142740
- See also: Caregiving in the U.S. 2009 Full Report — https://www.caregiving.org/research/open-data
- See also: U.S. Census Bureau QuickFacts — https://www.census.gov/quickfacts/TX